CLINICAL TRIAL: NCT03254836
Title: Sleep-wake Rhythm in the Perioperative Period in Patients Admitted for Elective Radical Surgery for Colorectal Cancer: an Observational Prospective Cohort Study.
Brief Title: Sleep and Survival in Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: Center of Surgical Science, Department of Surgery, Zealand University Hospital (Unknown)
Responsible Party: Principal Investigator, Michael Tvilling Madsen, M.D., Zealand University Hospital
Other Study IDs: MTM-V3; SJ-600 (Other: Region Zealand ethics Comittee)
Record Dates: First submitted 2017-08-15; First posted 2017-08-21 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Colorectal Neoplasm; Circadian Rhythm Sleep Disorder; Depression; Quality of Life; Sleep
Keywords: Actigraphy; Major Depression Inventory (MDI); Insomnia Severity Index (ISI)
MeSH Terms: conditions — Colorectal Neoplasms; Sleep Disorders, Circadian Rhythm; Depression | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal cancer undergoing elective surgery: All patients eligible for elective curative intended surgery for colonic adenocarcinoma at Zealand University Hospital.
  Patients will recieve treatment as per standard of care.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — Elective radical surgery for adenocarcinoma.

SUMMARY:
Objective The objective of the current trial is to investigate the effect of perioperative sleep and circadian rhythm on the natural course of survival among patient diagnosed with colorectal cancer. Concurrently, outcome measures like depression, fatigue, quality of life, and co-morbidity will be measured continuously in the short-, intermediate- and long-term period following diagnosis.

The a-priori hypothesis is that preoperative sleep and circadian disturbances is a prognostic marker of reduced overall survival. Likewise, preoperative sleep-wake disturbances at baseline are expected to result in overall universally reduced quality of life, increased depression and fatigue. Furthermore, development of sleep-wake disturbances in the postoperative period as compared to preoperative sleep-wake rhythm is expected to a prognostic marker of negative outcomes.

Target and study population The study population are all patients diagnosed with colorectal cancer in Region Zealand recruited consecutively from the trial initiation until study end each patient with an intended 5 year follow-up period. All available cases will be included in the trial.

Study design The study will be an observational prospective cohort study applying a longituditional repeated measure design.

Exposures and outcomes of interest The primary outcomes in the trial are sleep and circadian outcomes measured via actigraphy in the perioperative period.

Furthermore, cancer related survival and overall survival in the 5 year follow-up period is considered primary outcomes.

Secondary outcomes consist of consecutively measured depression, fatigue, quality of life, follow-up treatment and co-morbidity.

Exposure variables are primary related to the cancer, i.e. cancer stage, surgical treatment, oncological treatment, baseline co-morbidity and pharmacological treatment. Some of the secondary outcomes could be expected to serve as confounding or mediating factors.

Meaningful control for confounding will in the analysis phase be cancer stage and baseline sleep-wake rhythm status.

Sampling methods All available cases will be sought included in the trial. No formal sample size has been performed and continues inclusion into the trial will be performed during an 1,5 year period.

Statistical analyses The relationship between overall survival and baseline sleep-wake rhythm will be investigated using survival statistics and/or multivariate logistic regression.

Expected results The investigators expect to see a marked difference in overall survival among patients with sleep and circadian disturbances at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colorectal cancer as determined at the multi-disciplinary team conference.
* Admitted to elective radical surgery at the department of surgery at Zealand University Hospital
* Age above 18 years
* Informed consent

Exclusion Criteria:

* Non-ability to complete the study as assessed by the investigator
* Non-fluent in Danish.
* History of cognitive impairment (e.g. dementia)
* Paralysis or inability to answer study questioners electronically.
* Stadium 4 colonic adenocarcinoma with no surgical treatment options as determined at the multi-disciplinary conference.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients eligible for elective curative intended surgery for colonic or rectal adenocarcinoma at Zealand University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Actigraphy | Approximately 1 week preoperatively to 2 weeks postoperatively
  Assessment of activity using accelerometor - Sleep and circadian assesment.

SECONDARY OUTCOMES:
Major Depression Inventory | Baseline (approx. 1 week preoperatively), 2 weeks postoperatively, 3 months postoperatively, 6 months postoperatively, 12 months postoperativly, 24 months postoperatively, 36 months postoperatively, 60 months postoperatively.
  Assesment of depression
Insomnia Severity Index | Baseline (approx. 1 week preoperatively), 2 weeks postoperatively, 3 months postoperatively, 6 months postoperatively, 12 months postoperativly, 24 months postoperatively, 36 months postoperatively, 60 months postoperatively.
  Subjective sleep assesment
Quality of life assesment | Baseline (approx. 1 week preoperatively), 2 weeks postoperatively, 3 months postoperatively, 6 months postoperatively, 12 months postoperativly, 24 months postoperatively, 36 months postoperatively, 60 months postoperatively.
  EORCT-QLQ-C30
Quality of life assesment | Baseline (approx. 1 week preoperatively), 2 weeks postoperatively, 3 months postoperatively, 6 months postoperatively, 12 months postoperativly, 24 months postoperatively, 36 months postoperatively, 60 months postoperatively.
  EORCT-QLQ-CR29
Mortality | Baseline (approx. 1 week preoperatively), 2 weeks postoperatively, 3 months postoperatively, 6 months postoperatively, 12 months postoperativly, 24 months postoperatively, 36 months postoperatively, 60 months postoperatively.
  Baseline registration and follow-up assessments
Co-morbidity | Baseline (approx. 1 week preoperatively), 2 weeks postoperatively, 3 months postoperatively, 6 months postoperatively, 12 months postoperativly, 24 months postoperatively, 36 months postoperatively, 60 months postoperatively.
  Baseline registration and follow-up assessments
Drug prescription history (Drug name and dosage) | Baseline (approx. 1 week preoperatively), 2 weeks postoperatively, 3 months postoperatively, 6 months postoperatively, 12 months postoperativly, 24 months postoperatively, 36 months postoperatively, 60 months postoperatively.
  Baseline registration and follow-up assessments
Follow-up cancer treatment (Adjuvant chemotherapy, timing and duration) | Baseline (approx. 1 week preoperatively), 2 weeks postoperatively, 3 months postoperatively, 6 months postoperatively, 12 months postoperativly, 24 months postoperatively, 36 months postoperatively, 60 months postoperatively.
  Baseline registration and follow-up assessments

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Madsen, M.D., Principal Investigator — Department of Surgery, Zealand University Hospital
Locations (1):
- Department of Surgery, Zealand University Hospital, Roskilde, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Contact to study investigators avaliable at mitm@regionsjaelland.dk